CLINICAL TRIAL: NCT05306704
Title: High-Dose Vitamin D3 Supplementation in the Treatment of Human Immune Deficiency Virus Patients: A Double-Blind Randomized Control Trial
Brief Title: High-Dose Vitamin D3 Supplementation in the Treatment of Human Immune Deficiency Virus Patients Trial
Acronym: HDVDS-HIVT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of the Punjab (Other)
Collaborators: The National HIV/AIDS Programme (Other Government)
Responsible Party: Principal Investigator, Fatima Majeed, principal investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 12121218
Record Dates: First submitted 2021-04-21; First posted 2022-04-01 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: HIV-1-infection; Hypovitaminosis D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Olive Oil; 25-hydroxyvitamin D

STUDY DESIGN:
Intervention Model Description: Parallel group trial design. Parallel arm design is the most commonly used study design. In this design, subjects are randomized to one or more study arms and each study arm will be allocated a different intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Its double blind trail so trail is blinded for Participants, Care Provider, Investigator and Outcome Assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm: Olive oil (Placebo Comparator): In control arm participants will receive Placebo (Olive Oil) orally in all visits i.e from visit 1 to visit 4. Allocation of arms will be as per the pre-created random list.
  Interventions: Other: placebo Oil
- Vitamin-D (Active Comparator): In the Vitamin-D arm, participants will receive Vitamin-D (100000 IU) orally in all visits i.e from visit 1 to visit 4. Allocation of arms will be as per the pre-created random list.
  Interventions: Drug: 25-Hydroxyvitamin D

INTERVENTIONS:
Other: placebo Oil — participants will receive placebo(olive oil) orally in all visits from visit 1 to visit 4
  Other Names: Olive oil
  Arms: Control Arm: Olive oil
Drug: 25-Hydroxyvitamin D — Participants will receive vitamin D (100000IU) orally during all visits i.e. from visit-1 to visit-4
  Other Names: viatamin-D
  Arms: Vitamin-D

SUMMARY:
High-Dose Vitamin D3 in the Treatment of Human Immune Deficiency Virus Patients, A Double-Blind Randomized Control Trial Human immunodeficiency virus is a key challenge for global health. Vitamin D deficiency is common in people living with HIV infection. Antiretroviral therapy may create unique risk factors for vitamin D insufficiency, including alterations of vitamin D metabolism by ART.

DETAILED DESCRIPTION:
The study is designed to evaluate the effect of high dose Vitamin-D supplementation in the treatment of HIV patients with Antiretroviral therapy.

Furthermore, in secondary outcomes study will evaluate the effects of high dose vitamin-D supplementation by Pre & Post assessments of CD4 count and PCR count.

Secondary outcomes also includes the effects of high dose vitamin-D supplementation by Pre & Post assessments of SGPT, SGOT, ALP and Bilirubin.

Tertiary outcomes includes the effects of high dose vitamin-D supplementation by Pre & Post assessments of Hb, Lymphocytes, Monocytes, Eosinophil, Platelet count and Basophil count.

A sample size of 95 patients were recruited in Said Mitha Teaching Hospital Lahore.

Study is planned in two groups including 1) ARV + Vitamin-D3 2) ARV + Placebo. Methods/design: A randomized placebo controlled double-blind clinical trial of patients with age 19-50 years.

The primary outcome will be assessed by analyzing the difference change in the Vitamin-D Levels from Day 1 to Week 12. Secondary outcomes including viral load count, CD4 count, elevated levels of LFTs, will also be assessed by analyzing the mean difference in their values on week 12 after the supplementation of high dose Vitamin-D. Tertiary outcomes (Hematology) including Hb, HCT, TLC, Eosinophil's count, Neutrophils count, Monocytes and Platelets Data will be collected on a predefined Performa. All information will be entered in SPSS for the analysis.

Discussion: High dose Vitamin D supplementation in HIV-infected patients has not been previously investigated in Pakistan and it is unknown whether increasing levels is associated with improved clinical outcome or not. Therefore, it is significant to conduct a study to know the effect of vitamin D in the treatment of HIV patients with antiretroviral therapy.

Keywords: AIDS, HIV, anti-retroviral therapy, high dose 25-hydroxy Vitamin-D level, CD4 count, viral load.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 19 years and above
2. Vitamin-D levels less than 20ng/ml
3. Not taking any kind of Vitamin-D supplementation or Mega Doses for last six months
4. Written Informed Consent Form
5. PCR Positive Patients

Exclusion Criteria:

1. Pregnant and Lactating Women
2. Ability to take Study Medication Orally

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Primary Outcome is to achieve normal physiological level by Vitaman-D3 supplementation in HIV positive patients | Within 12 Weeks
  Optimal level of Vitamin-D3 i.e >20ng/ml in HIV patients

SECONDARY OUTCOMES:
The secondary outcome is to assess the mean differences in CD4 count | Within 12 Weeks
  Optimal value of CD4 count is 500-1500 cells/mm3 the unit of CD4 count is cells/mm3
To measure the effect of our intervention on PCR value copies/µL. | within 12 weeks
  PCR normal value is usually comes under detected and non-detected category and its unit is copies/µL
To measure the effect of intervention on the viral load value | within 12 weeks
  The normal value of viral load must be zero and measures in copies/µL of the blood.
To measure the effect of intervention on SGPT | Within 12 weeks
  The normal value of SGPT is measured in (µL)
To measure the effect of intervention on SGOT | Within 12 weeks
  The normal value of SGOT is measured in (µL)
To measure the effect of intervention on ALP | Within 12 weeks
  The normal value of ALP is measured in (µ/l)
To measure the effect of intervention on Bilirubin | Within 12 weeks
  The normal value of Bilirubin measured in (mg/dl)

OTHER OUTCOMES:
To access the effect of the intervention on Lymphocytes | within 12 weeks
  The units for Lymphocytes is in percentage %
To access the effect of intervention on Monocytes | within 12 weeks
  The units for Monocytes is in percentage %
To access the effect of intervention on Hemoglobin | within 12 weeks
  The hemoglobin level is measured in g/dl
To access the effect of the intervention on Platelets count | Within 12 weeks.
  The platelets count is normally measured in 1000/µL
To access the effect of the intervention on Eosionophil | Within 12 weeks
  The platelets count is normally measured in percentage %
To access the effect of the intervention on Basophil | Within 12 weeks
  The Basophil count is normally measured in percentage %

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Govt Said Mitha Teaching Hospital Lahore, Lahore, Punjab/ lahore/Pakistan
  - Fatima Majeed, Lahore, Punjab/ lahore/Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT05306704/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT05306704/SAP_001.pdf
  • Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT05306704/ICF_002.pdf